CLINICAL TRIAL: NCT05037656
Title: University of Guam/University of Hawaii Cancer Center Partnership for Cancer Health Equity, Full Project I: Developing and Testing a School-Based Curriculum for E-cigarette, Tobacco, and Betel (Areca) Nut Use Prevention for Guam Youths
Brief Title: Testing a School-Based E-cigarette, Tobacco, and Betel (Areca) Nut Use Prevention Curriculum for Guam Youths
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guam (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Hawaii Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2U54CA143728-11 (NIH); U54CA143728 (NIH)
Record Dates: First submitted 2021-07-30; First posted 2021-09-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Smoking; Vaping; Tobacco Chewing
Keywords: tobacco; e-cigarette; Areca nut; Prevention; Adolescents
MeSH Terms: conditions — Tobacco Smoking; Vaping; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Students in the control group will receive the standard health education curriculum.
- Experimental (Experimental): Students in the treatment group will receive the school-based classroom curriculum.
  Interventions: Behavioral: School-based curriculum

INTERVENTIONS:
Behavioral: School-based curriculum — Participants will be randomized, at the school level, to receive either the e-cigarette/tobacco/areca nut use prevention curriculum or the standard of care (i.e., control). The curriculum will be implemented using 5 intensive in-class lessons over the span of 6 weeks. All sessions of the curriculum follow the same basic format: a) an introduction and/or review of the past lesson, b) a cultural wall activity, c) a video, d) 1-2 interactive activities, and e) a wrap-up activity. Lessons are designed such as to help improve knowledge about drugs and correct cognitive misperceptions and to train on skills to resist normative social influence. Participants will complete identical survey questionnaires for assessments at 3 time-points: pretest (baseline, before implementing the intervention), immediate posttest (following the end of the intervention), and six-month follow-up. The surveys will be administered in the classroom, during regular school hours.
  Arms: Experimental

SUMMARY:
The people of the U.S. Affiliated Pacific Islands (USAPI) face higher cancer incidence, especially lung/bronchia and head-and-neck cancer, and poorer cancer outcomes, compared with the U.S. nationally. This may partly be driven by the high rates of cigarette smoking and betel (areca) nut use in the USAPI. Previous data suggest that that adolescents on Guam, as young as middle school students report markedly higher e-cigarette and tobacco product use prevalence in the USAPI compared with the USAPI nationally. Guam youths are also at risk for the use of betel nuts. Yet, currently there are no tobacco product/areca nut use prevention programs that have been developed for and tested specifically USAPI adolescents. The proposed study will develop a school-based substance use prevention curriculum for e-cigarette, tobacco product, and areca nut use prevention among Guam youths. The curriculum will use lessons incorporating innovative videos and culturally grounded activities.

The study's specific aims are:

1. To develop a school-based curriculum for e-cigarette, tobacco product (i.e., cigarette, smokeless tobacco), and betel nut use prevention among middle school students in Guam.
2. Test the efficacy of the school-based curriculum in a randomized controlled trial.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

The study focuses on e-cigarette, tobacco and areca nut prevention among adolescents in Guam. By developing and testing a school-based e-cigarette, tobacco and areca nut prevention program, the project will target psychosocial, lifestyle, and environmental/physical factors contributing to cancer disparities in the US Affiliated Pacific Islands (USAPI). Thus far, nationally, there has been limited effort in terms of developing a theoretical framework that would attempt to explain tobacco and areca nut use etiology among USAPI youth. Previous research indicates that social and environmental influences play key roles in shaping tobacco and areca nut use among USAPI youths. In addition, skills needed to resist social influence appear to be protective against tobacco and areca nut use. Particularly, past research has found peer influence and environmental risk factors such as parental permissiveness, ease of access to tobacco/areca nut at home and school and through adults and friends, to be strongly associated with current tobacco/areca nut use. On the other hand, competence in navigating through social situations conducive to tobacco/areca nut use and refusal self-efficacy (i.e., confidence in being able to say "no" at the face of peer pressure) have been found to be strongly associated with lower likelihood of current tobacco/areca nut use.

The curriculum to be developed and tested will focus on informing adolescents on the risks of tobacco product/areca nut use as well as training adolescents on social influence resistance skills in a culturally appropriate way, using innovative use of video vignettes. The intervention will seek to influence behavior (i.e., prevention and reduction of tobacco product/areca nut use) by countering the cognitive predispositions to tobacco product/areca nut use (e.g., by increasing risk perceptions, reducing positive expectancies) and by providing youths with skills to resist specific social influence to use tobacco products/areca nut on specific occasions.

RESEARCH DESIGN

This is an experimental study. Of the eight public middle schools in Guam, four schools will be randomly assigned to the "Treatment" and four to the "Control" condition. Students in the Treatment schools will receive the classroom-based curriculum whereas students in the Control schools will receive the standard health education curriculum (treatment-as-usual). Participants will be assessed at pre-test, immediate post-test, and six months after the post-test. Note that the decision to provide an intervention, albeit weaker, to the control group was guided by the ethics of good community practice. In preliminary discussions with schools, principals unanimously expected an intervention.

Participants

Participants will be 600 Guam middle school students. Based on a pilot study, the mean age of the participants is likely to be 12.7 years (SD = .89); 49% of the participants are likely to be girls; and 47% of the participants are likely to be Chamorus, 27% other Pacific Islanders, and 25% non-Pacific Islanders (i.e., Filipinos, Chinese, Japanese, white, and others). Treatment and Control conditions will represent roughly equal proportion of participants.

Recruitment

All eight public middle schools will be involved in the study. The Guam Department of Education (GDOE) has been very supportive of this study. At each school, seven classes will be randomly selected to participate in the study.

Intervention delivery

The classroom curriculum will begin in the Treatment schools within two weeks of the pre-test. The social media campaign will begin in all schools around the same time. Below we provide details on the delivery of each intervention component.

Classroom-based curriculum: Curriculum implementation. The curriculum will be delivered by teachers of the Treatment schools who normally teach physical health education classes. The curriculum will be implemented once a week for 45-60 minutes over a 10-week academic quarter in a required physical/health education course. All sessions of the curriculum will follow the same basic format of Ho'ouna Pono. Each lesson will be aligned with the Guam Content and Performance Standards for Health (6-8 grade) and/or the National Common Core Standards in public education. The teachers will be trained to implement the curriculum through a hybrid (i.e., in-person and virtual), credit-granting course sanctioned through the GDOE.

Data collection

Data will be collected at three timepoints from students in both Treatment and Control conditions: pre-test (baseline), immediate post-test (i.e., approximately a week after the last classroom-based curriculum session is delivered), and six months after the post-test. Data will be collected using self-report questionnaires, although self-report of cigarette use and areca nut use will also be validated using biochemical verification methods in random subsample of participants. At each timepoint the same questionnaire will be administered across Treatment and Control groups. The self-report questionnaire will include the following assessment measures.

Measures

Demographic measures. Age, gender, socio-economic status, and ethnicity will be assessed. Socio-economic status (SES) is measured based on participants' report on their parents' level of education. However, past research shows that a good proportion of adolescents do not know about parental education level. Hence, a measure of household crowdedness (i.e., the number of usual residents in a household divided by the number of rooms in the house) will also be included to assess SES. Ethnicity will be assessed with a single item previously used by us in Guam. A measure of acculturation will also be included.

Intrapersonal/Dispositional variables. These will include self-control, assessed in terms of behavioral and emotional self-control; sensation seeking; social competence in resisting social influence; general self-efficacy; refusal self-efficacy; and self-esteem. The items specific to substance use will be adapted for cigarette smoking, e-cigarette use, chewing tobacco use, and areca nut use.

Social/Interpersonal variables. These will include family and friend areca nut/tobacco product use, perceived norms, and social normative beliefs. Perceived norms and social normative beliefs will be adapted for cigarette smoking, e-cigarette use, chewing tobacco use, and areca nut use.

Cultural/Environmental variables. These will include availability of areca nut/tobacco at home and school, parental permissiveness, knowledge about areca nut/tobacco products, areca nut/tobacco product use expectancies, and areca nut/tobacco product use harm/risk perceptions.

Exposure to content relevant to tobacco products and areca nut on social media. Exposure will be assessed using 12 items previously validated by us for tobacco products and areca nut. The items assess exposure to user-generated content, traditional marketing, and prevention messages.

Areca nut and tobacco product use susceptibility. Areca nut use and tobacco product use susceptibility will be separately assessed for cigarette smoking, e-cigarette use, chewing tobacco use, and areca nut use with a measure of adolescent substance use intentions (13), adapted for each substance.

Areca nut and tobacco product use. The study will assess areca nut only use, combined areca nut and tobacco use, cigarette smoking, e-cigarette use, and chewing tobacco use separately. For each of these substance use outcomes, the study will assess lifetime (ever) use (e.g., "Have you ever used a areca nut in your lifetime?") and past-30-day use (e.g., "In the past 30 days, on how many days did you use areca nut?). Self-report measures of adolescent substance use have been extensively studied for their validity, by using multiple methods, and they have consistently been found to be valid.

Data Analysis

Data analysis will be performed with the help of the PIPCHE Biostatistics Core. The primary goal of the analysis is to examine the efficacy of this group randomized trial (16) for substance use prevention among middle schoolers. Aim 1 will compare the change in tobacco and areca nut beliefs, attitudes, initiation and use over time between the two randomization conditions, accounting for the clustering of classes within schools and the randomization unit of schools. In particular, the following mixed regression will be performed: where Z is a vector of covariates for each student at each time point, T is time, G is randomization group, TxG is the interaction of time and group, and η is a random effect for clustering of classes within schools and δ is a random effect for repeated measures within student. The link function ƒ is linear for continuous outcomes, such as a belief score, and logistic for dichotomous outcomes, such as initiation; outcomes will be transformed as needed to meet model assumptions. Potential covariates would include age, sex of student, grade, ethnicity, parent's education level, sensation seeking and teacher sex. Time T will be parameterized as indicator variables for baseline, post-intervention, and six month follow-up, or as continuous months if warranted by a monotonic change over time. The intervention effect will be assessed by the F-test in linear models and chi-square test in logistic models for the βTG parameter, with the degrees of freedom adjusted to account for the eight randomization units. Covariate-adjusted means and 95% confidence intervals will be estimated from the models for each level of randomization group and time point. The SAS procedure GLIMMIX will be used to fit these mixed models, which can accommodate data from students with missing data at some time points and allow for the results to be more generalizable to the student population. However, the study will assess the effect of missing data by comparing characteristics of students with complete and incomplete data and will perform multiple imputation if needed. As exploratory analyses, the study will test for differential intervention effects in subgroups, such as defined by student ethnicity, by adding interaction terms between subgroup and treatment/time variables and assessing the significance of the three way interaction. The study will also explore the effect of dose of the intervention, by studying change in outcomes by number of session attended among students in the intervention schools, and the effect of fidelity assessments of the intervention per classroom.

Statistical Power

The sample size of eight schools, with four randomized to each condition, each with seven classes of 20 students, is sufficient to ensure adequate statistical power to detect meaningful differences between intervention arms in all outcomes. For Aim 1, the effect size, Cohen's d was calculated based on a z-test comparing means and a chi-square test comparing proportions, with n=8 schools, with four schools per randomization condition, each with 20 students. The variance of the differences was adjusted for the Design Effect of the present study, accounting for the clustering in a group-randomized trial (GRT) by adjusting the test degrees of freedom to the number of communities. The intraclass correlation coefficient (ICC) of outcomes within schools and within class in schools was set to 0.01-0.02, based on past school-based studies, for an overall ICC varying between 0.02 to 0.04. The study assumed a critical level α of 0.05 (two-sided) or 0.005 (Bonferroni-corrected for 10 tests), a power of 80%, and up to a 20% attrition in sample size at post-intervention. The effect size for a test of means is medium at 0.29-0.38 for α=0.05 and at 0.37-0.50 for α=0.005. The following differences between conditions in changes in proportions will be detectable with α=0.05: 0% versus 4.0% and 3% versus 10.5%; and with α=0.005: 0% versus 6.5% and 3% versus 15.5%.

ELIGIBILITY:
Inclusion Criteria:

* All students enrolled in public middle schools in Guam (age: 11-15 years old)
* Provide signed parental informed consent and student assent

Exclusion Criteria:

* Participants whose parents decline participation or students who decline participation.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 538 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Youth Risk Behavior Surveillance (YRBS) Survey-based self-reported past-30-day tobacco, e-cigarette, and areca nut use | Outcomes will be assessed at baseline (pre-test), 5 weeks after baseline, immediately following curriculum/standard of care delivery (i.e., post-test), and 6 months after baseline (follow-up)
  Tobacco, e-cigarette, and areca nut use behavior will be assessed using a standardized self-report measure of recent use that is use in the national YRBS survey. The questionnaire item will ask: "In the past 30 days, on how many days did you smoke a cigarette?" This question will be adapted for e-cigarette and areca nut. Response options include: "0 days," "1-2 days," "3-5 days," "6-9 days," "10-19 days," "20-29 days," "all 30 days."
Changes in Pierce's Smoking Susceptibility Scale (also adapted for e-cigarette and areca nut use) | Outcomes will be assessed at baseline (pre-test), 5 weeks after baseline, immediately following curriculum/standard of care delivery (i.e., post-test), and 6 months after baseline (follow-up)
  This is a standardized self-report measure containing 4 items originally designed to assess smoking susceptibility among adolescents. In addition to the original measure, the current study will also adapt the measure to assess e-cigarette and areca nut use susceptibility. The 4 items are: "Do you think you will smoke a cigarette soon?", "Do you think you will smoke a cigarette in the next year?", "Do you think in the future you might experiment with cigarettes?", "If one of you friends were to offer you a cigarette, would you smoke it?"

SECONDARY OUTCOMES:
Kendall Wilcox Self-control Scale | Outcomes will be assessed at baseline (pre-test), 5 weeks after baseline, immediately following curriculum/standard of care delivery (i.e., post-test), and 6 months after baseline (follow-up)
  This is a standardized self-report scale containing 7 items designed to assess generalized self-control, including impulsivity and behavioral self-control.
Jackson et al.'s Social Competence Scale | Outcomes will be assessed at baseline (pre-test), 5 weeks after baseline, immediately following curriculum/standard of care delivery (i.e., post-test), and 6 months after baseline (follow-up)
  This is a standardized self-report scale containing 27 items designed to assess social competence is resisting social influence related to tobacco and other substance use among adolescents.
Sherer et al.'s General Self-Efficacy Scale | Outcomes will be assessed at baseline (pre-test), 5 weeks after baseline, immediately following curriculum/standard of care delivery (i.e., post-test), and 6 months after baseline (follow-up)
  This is a standardized self-report scale containing 6 items designed to assess confidence in performing a behavior. Sample items include "When I make plans, I am certain I can make them work", "If I can't do a job the first time, I keep trying until I can", and "When I have something unpleasant to do, I stick to it until I finish it".
Flay et al.'s Refusal Self-Efficacy | Outcomes will be assessed at baseline (pre-test), 5 weeks after baseline, immediately following curriculum/standard of care delivery (i.e., post-test), and 6 months after baseline (follow-up)
  This is a standardized self-report scale containing 6 items designed to assess confidence in refusing tobacco and other substance use offers.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Dalisay, PhD, Principal Investigator — University of Guam; Pallav Pohkrel, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- Guam Department of Education, Tiyan, Guam, Guam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okamoto SK, Helm S, Ostrowski LK, Flood L. The Validation of a School-Based, Culturally Grounded Drug Prevention Curriculum for Rural Hawaiian Youth. Health Promot Pract. 2018 May;19(3):369-376. doi: 10.1177/1524839917704210. Epub 2017 Apr 26. PMID 28443350
- [Background] Okamoto SK, Helm S, Chin SK, Hata J, Hata E, Okamura KH. The implementation of a culturally grounded, school-based, drug prevention curriculum in rural Hawai'i. J Community Psychol. 2020 May;48(4):1085-1099. doi: 10.1002/jcop.22222. Epub 2019 Jul 23. PMID 31332808
- [Background] Okamoto SK, Helm S, McClain LL, Dinson AL. The development of videos in culturally grounded drug prevention for rural native Hawaiian youth. J Prim Prev. 2012 Dec;33(5-6):259-69. doi: 10.1007/s10935-012-0281-0. PMID 23143071
- [Background] Flay BR. The promise of long-term effectiveness of school-based smoking prevention programs: a critical review of reviews. Tob Induc Dis. 2009 Mar 26;5(1):7. doi: 10.1186/1617-9625-5-7. PMID 19323827
- [Background] Pokhrel P, Sussman S, Stacy A. Relative effects of social self-control, sensation seeking, and impulsivity on future cigarette use in a sample of high-risk adolescents. Subst Use Misuse. 2014 Mar;49(4):343-51. doi: 10.3109/10826084.2013.841241. Epub 2013 Oct 4. PMID 24093522
- [Background] Okamoto SK, Helm S, Pel S, McClain LL, Hill AP, Hayashida JK. Developing empirically based, culturally grounded drug prevention interventions for indigenous youth populations. J Behav Health Serv Res. 2014 Jan;41(1):8-19. doi: 10.1007/s11414-012-9304-0. PMID 23188485
- [Background] Herzog TA, Murphy KL, Little MA, Suguitan GS, Pokhrel P, Kawamoto CT. The Betel Quid Dependence Scale: replication and extension in a Guamanian sample. Drug Alcohol Depend. 2014 May 1;138:154-60. doi: 10.1016/j.drugalcdep.2014.02.022. Epub 2014 Feb 26. PMID 24629627
- [Background] Moss J, Kawamoto C, Pokhrel P, Paulino Y, Herzog T. Developing a Betel Quid Cessation Program on the Island of Guam. Pac Asia Inq. 2015 Fall;6(1):144-150. PMID 27057560
- [Background] Dalisay F, Buente W, Benitez C, Herzog TA, Pokhrel P. Adolescent betel nut use in Guam: beliefs, attitudes and social norms. Addict Res Theory. 2019;27(5):394-404. doi: 10.1080/16066359.2018.1538410. Epub 2019 Jan 11. PMID 31231175
- [Background] Gentzke AS, Creamer M, Cullen KA, Ambrose BK, Willis G, Jamal A, King BA. Vital Signs: Tobacco Product Use Among Middle and High School Students - United States, 2011-2018. MMWR Morb Mortal Wkly Rep. 2019 Feb 15;68(6):157-164. doi: 10.15585/mmwr.mm6806e1. PMID 30763302
- [Background] Oakley E, Demaine L, Warnakulasuriya S. Areca (betel) nut chewing habit among high-school children in the Commonwealth of the Northern Mariana Islands (Micronesia). Bull World Health Organ. 2005 Sep;83(9):656-60. Epub 2005 Sep 30. PMID 16211156
- [Background] Milgrom P, Tut OK, Gilmatam J, Gallen M, Chi DL. Areca use among adolescents in Yap and Pohnpei, the Federated States of Micronesia. Harm Reduct J. 2013 Oct 17;10:26. doi: 10.1186/1477-7517-10-26. PMID 24134714
- [Background] Paulino YC, Novotny R, Miller MJ, Murphy SP. Areca (Betel) Nut Chewing Practices in Micronesian Populations. Hawaii J Public Health. 2011 Mar;3(1):19-29. PMID 25678943
- [Background] Soneji S, Barrington-Trimis JL, Wills TA, Leventhal AM, Unger JB, Gibson LA, Yang J, Primack BA, Andrews JA, Miech RA, Spindle TR, Dick DM, Eissenberg T, Hornik RC, Dang R, Sargent JD. Association Between Initial Use of e-Cigarettes and Subsequent Cigarette Smoking Among Adolescents and Young Adults: A Systematic Review and Meta-analysis. JAMA Pediatr. 2017 Aug 1;171(8):788-797. doi: 10.1001/jamapediatrics.2017.1488. PMID 28654986
- [Background] Buente W, Dalisay F, Pokhrel P, Kramer HK, Pagano I. An Instagram-Based Study to Understand Betel Nut Use Culture in Micronesia: Exploratory Content Analysis. J Med Internet Res. 2020 Jul 9;22(7):e13954. doi: 10.2196/13954. PMID 32673220
- [Background] Pierce JP, Choi WS, Gilpin EA, Farkas AJ, Berry CC. Tobacco industry promotion of cigarettes and adolescent smoking. JAMA. 1998 Feb 18;279(7):511-5. doi: 10.1001/jama.279.7.511. PMID 9480360
- [Background] Wills TA, Bantum EO, Pokhrel P, Maddock JE, Ainette MG, Morehouse E, Fenster B. A dual-process model of early substance use: tests in two diverse populations of adolescents. Health Psychol. 2013 May;32(5):533-42. doi: 10.1037/a0027634. PMID 23646836
- [Background] Jackson C, Henriksen L, Dickinson D, Levine DW. The early use of alcohol and tobacco: its relation to children's competence and parents' behavior. Am J Public Health. 1997 Mar;87(3):359-64. doi: 10.2105/ajph.87.3.359. PMID 9096534
- [Background] Sherer M, Mercandante JEMB, Prentice-Dunn S, Jacobs B, Rogers RW. The self-efficacy scale: construction and validation. Psychological Reports. 1982;51(2):663-71.
- [Background] Flay BR, Hu FB, Siddiqui O, Day LE, Hedeker D, Petraitis J, Richardson J, Sussman S. Differential influence of parental smoking and friends' smoking on adolescent initiation and escalation of smoking. J Health Soc Behav. 1994 Sep;35(3):248-65. PMID 7983337